CLINICAL TRIAL: NCT04401670
Title: Cervical Cancer Screening Strategies in Women Living With HIV and HIV Uninfected Women in Cameroon
Brief Title: Cervical Cancer Screening in Cameroon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Adebola Adedimeji, Research Associate Professor, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2016-6070; 3P30CA013330 (NIH)
Record Dates: First submitted 2020-05-18; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Cervical Cancer; HIV/AIDS
Keywords: HIV; HPV screening; cervical cancer; self sampling; human papillomavirus
MeSH Terms: conditions — Uterine Cervical Neoplasms; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Masking Description: The US pathologist was masked to the original cytologic interpretation but unmasked to being hrHPV positive to reduce influence of how the slides were read.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triage with different options (Other): * Self-Collection: hrHPV and Biomarkers Testing (among hrHPV+)
  * ThinPrep Specimen: Liquid-Based Cytology (LBC), hrHPV Testing, and Biomarker Testing (among hrHPV+)
  * Visual Inspection after Acetic Acid (VIA)
  Interventions: Other: HPV screening and triage tests; Behavioral: HPV self-sampling

INTERVENTIONS:
Other: HPV screening and triage tests — The participants underwent a pelvic exam to have a provider-collected sample placed in PreservCyt [Hologic, Inc., Bedford, MA, USA] and a visual inspection by acetic acid (VIA) by a nurse.
Behavioral: HPV self-sampling — The participant was escorted by the nurse to a private room and given instructions on how to self-collect their sample using "Just for Me" sampler [Preventive Oncology International, Cleveland, OH, USA].

SUMMARY:
Human immunodeficiency virus-infected (HIV[+]) women have a several-fold increased risk of invasive cervical cancer (ICC) as well as increased risk of cervical pre-cancer. In low- and middle-income countries (LMICs), ICC is the 1st or 2nd most common cause of cancer and cancer-related death in women. Rates of ICC and ICC-related mortality are particularly high in Sub-Saharan Africa, which also has the highest rates of HIV infection in the world. Although prophylactic HPV vaccines may be the optimal cervical cancer prevention strategy, 2-3 generations of at-risk HIV[+] and HIV[-] women are already highly exposed to human papillomavirus (HPV) and would not benefit from (and will not be immunized with) HPV vaccine. Thus cervical cancer screening is needed for the foreseeable future. However, Pap testing is expensive and requires a complex clinical and lab infrastructure that does not generally exist in LMICs; strategies based on high-risk HPV (hrHPV) testing or visual inspection after acetic acid (VIA) are promising but are either too non-specific, leading to over-referral for colposcopy or over-treatment, or are too insensitive, respectively. Thus, inexpensive, easily implemented, and effective cervical cancer screening methods are greatly needed in Sub-Saharan Africa, especially for HIV[+] women. This cervical cancer screening study of 1,200 women (800 HIV[+] and 400 HIV[-] women), aged 25-59 years, living in Cameroon, utilized our existing research site. The investigators evaluated screening tests (hrHPV testing, VIA and Pap), traditional triage tests (HPV16/18/45 detection, VIA, Pap), and promising new biomarkers for triage (Ki-C67, TOP2a, CDKN2A, and HPV viral load) of screen-positive women. All screen positives underwent rigorous disease ascertainment to obtain unbiased estimates of sensitivity, specificity, and positive and negative predictive value. The goal of this study was to establish the foundation and capacity for future studies designed to reduce the burden of HPV-associated cancers in the Cameroon population. It will inform Cameroon and other countries with high HIV burdens on the best strategies for cervical cancer screening in their HIV[+] and HIV[-] women.

ELIGIBILITY:
Inclusion Criteria:

* Women living in Limbe town and neighborhood
* Confirmed to be HIV[+] or HIV[-]
* Have never undergone cervical cancer screening, with no history of ICC
* Willing and able to competently understand and provide written, informed paper-based consent
* Women who are having a menstrual period will be deferred for 2 weeks from participating in the study

Exclusion Criteria:

* Pregnant women
* Women with signs of abnormalities
* Non-menstrual bleeding suggestive of ICC
* Without a cervix because they have undergone hysterectomy
* Based on the judgment of the clinicians not sufficiently healthy to participate in a research study

Ages: 25 Years to 56 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 873 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Triage Testing of HIV[+] and HIV[-] Women for Detection of CIN2+ and CIN3+ | 0 days
  To evaluate and compare the clinical performance of high-risk human papillomavirus (hrHPV) DNA testing using provider-collected specimens (Provider/hrHPV) and self-collected specimens (Self/hrHPV), visual inspection after acetic acid (VIA), and liquid-based cytology (LBC) for detection of cervical intraepithelial neoplasia (CIN) grade 2 or more severe diagnoses (CIN2+) and grade 3 or more severe diagnoses (CIN3+) in HIV[+] and HIV[-] women.
Triage Testing of HPV-Positive Women for the Detection of CIN2+ and CIN3+ | 0 days
  To compare the clinical performance of VIA, detection of the most carcinogenic hrHPV genotypes HPV16, 18, or/and 45, and biomarkers Ki-67, p16INK4a, and TOP2A mRNA, HPV viral load, and LBC as triage strategies for hrHPV-positive women for detection of CIN2+ and CIN3+.
Age-Specific Prevalence of Screen Positives in Limbé | 0 days
  To measure the age-group specific prevalence of hrHPV DNA, LBC, and VIA positivity, and CIN2+ and CIN3+ in HIV[+] and HIV[-] women living in Limbé, Cameroon.

SECONDARY OUTCOMES:
Qualitative interviews to assess acceptability and feasibility of self-collection from women | 0 days
  To identify micro- and meso-level factors from an exploratory qualitative analysis using data obtained through focus group discussions and in-depth interviews to evaluate acceptability and feasibility of self-sampling for hrHPV testing among HIV[+] and HIV[-] women living in Limbé, Cameroon. This approach was used to better understand and describe women's knowledge, attitudes, and practices regarding cancers in general, cervical cancer, HPV infection, screening as well as behavioral and structural facilitators and barriers to cervical cancer prevention. Additional information was obtained to assess and compare perceptions and preferences for self-versus health provider-collected biological specimens to understand women's preferences given peculiar contextual factors that facilitate or inhibit access to cervical cancer screening for women at risk.

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Castle, Principal Investigator — Albert Einstein College of Medicine; Adebola Adedimeji, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Limbé Regional Hospital, Limbe, Cameroon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castle PE, Ajeh R, Dzudie A, Kendowo E, Fuhngwa N, Simo-Wambo AG, Nsame D, Orock E, Hebert TM, Pierz AJ, Murokora D, Anastos K, Adedimeji A. A comparison of screening tests for detection of high-grade cervical abnormalities in women living with HIV from Cameroon. Infect Agent Cancer. 2020 Jul 11;15:45. doi: 10.1186/s13027-020-00311-w. eCollection 2020. PMID 32676125